CLINICAL TRIAL: NCT01473498
Title: Personalized Haemodynamic Management of Septic Shock: Influence of Mean Arterial Pressure Level on Renal Function: Randomized Controlled Trial
Brief Title: Personalized Mean Arterial Pressure Management on Renal Function During Septic Shock
Acronym: DORESEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P091103
Record Dates: First submitted 2011-10-14; First posted 2011-11-17 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Septic Shock; Acute Kidney Injury
Keywords: Sepsis; Acute kidney injury; Mean arterial pressure; Catecholamines; Renal doppler
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test group (Experimental): Patients will be treated with fluid and norepinephrine to achieve and maintain a mean arterial pressure of 65 mm Hg. Then they will be randomized in two groups.
  In the first group (study group, n=30), mean arterial pressure will be increased to 85 mm Hg for 72 hours by increasing the dose of norepinephrine in patients (A maximum dose of 1.2 mcg / kg / min is not exceeded). Key details, e.g., for drugs include dosage form, dosage, frequency and duration.
  Interventions: Other: Haemodynamic management
- Control group (Active Comparator): Patients will be treated with fluid and norepinephrine to achieve and maintain a mean arterial pressure of 65 mm Hg. Then they will be randomized in two groups.
  In this group (control group, n=30), mean arterial pressure will be maintained at 65 mm Hg.
  Interventions: Other: Haemodynamic management

INTERVENTIONS:
Other: Haemodynamic management — Patients will be treated with fluid and norepinephrine to achieve and maintain a mean arterial pressure of 65 mm Hg. Then they will be randomized in two groups.
  In the first group (study group, n=30), mean arterial pressure will be increased to 85 mm Hg for 72 hours by increasing the dose of norepinephrine in patients.
  Arms: Control group
Other: Haemodynamic management — Patients will be treated with fluid and norepinephrine to achieve and maintain a mean arterial pressure of 65 mm Hg. Then they will be randomized in two groups.
  In this group (control group, n=30), mean arterial pressure will be maintained at 65 mm Hg.
  Arms: Test group

SUMMARY:
Sepsis is the most severe complication of infections. Sepsis-associated Acute kidney injury (AKI) is commonly encountered in critically ill patients and independently predicts poor outcome. Unfortunately, no drug or management strategy was able to reduce incidence of AKI. To adapt the level of mean arterial pressure according to local renal hemodynamic evaluated by renal Doppler could lead to a better renal perfusion, and then less AKI.

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is a frequent and serious complication of sepsis. Renal ischemia plays a major role in the pathophysiology of sepsis-associated AKI. There is currently no treatment to prevent or to treat AKI. It has been shown that a resistivity index (RI) greater than 0.74 of patients with septic shock could predict the occurrence of renal failure, and that increase mean arterial pressure (MAP) with norepinephrine could decrease RI. Hence, we propose to compare the frequency and the severity of the sepsis-associated AKI according to the early hemodynamic management of septic shock. Patients will be randomized in a classic group (MAP 65 mmHg) and an interventional group (MAP 85 mmHg). We can thus determine whether the level of MAP influences renal function, and whether this influence of MAP is dependent of renal perfusion assessed by renal Doppler.

Participants will be followed for the duration of hospital stay, an expected average of 4 weeks.

Primary endpoint:

-Presence and severity of sepsis-associated AKI at day 7.

Secondary endpoints:

* Acute renal failure measured by Classification AKI at day 28.
* Acute renal failure as measured by the RIFLE classification in the fourth to seventh day and 28th day.
* Use of renal replacement therapy during hospitalization in intensive care unit
* Mortality at day 28 Duration of study: Recruitment: 10 months, the patient monitoring: 28 days ± 3 days, total test duration: 11 months

ELIGIBILITY:
Inclusion Criteria:

* Any patient with septic shock may be included in the next 6 to 16h
* Age > 18 years old and <= 80 years

Exclusion Criteria:

* Chronic renal failure (Baseline serum creatinine > 120 mmol/L)
* Chronic cardiac failure (Left ventricle ejection fraction < 40%)
* Pregnancy
* Urinary Tract Infection
* Patients with a left ventricular dysfunction ( ventricular ejection fraction <40%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury according to RIFLE score | at 7 days

SECONDARY OUTCOMES:
Need for renal replacement therapy | during hospitalization
  including metabolic indications (Azotemia Serum urea ≥ 36mmol/L (100 mg/dL) ; Uremic complications : encephalopathy, pericarditis, bleeding ; Hyperkalemia K+ ≥ 6 mmol/L and/or electrocardiogram abnormalities ; Hypermagnesemia ≥4 mmol/L and/or anuria/absent deep tendon reflexes ; Acidosis Serum pH ≤ 7.15), Oligo-anuria Urine output <200mL/12 h or anuria, Fluid overload like Diuretic-resistant organ edema in the presence of acute kidney injury.
All cause mortality | at 28 days
  All Cause mortality at 28 days, including refractory shock, refractory hypoxia, multiple organ failure, decisions to forgo life-sustaining therapies (DFLSTs)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DURANTEAU, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Reanimation Chirurgicale - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre, France